CLINICAL TRIAL: NCT00297648
Title: A Phase IIIB Multicentre Open Label 54 Weeks Clinical Trial Evaluating Certolizumab Pegol, a PEGylated Fab Fragment of Humanized Antibody to Tumor Necrosis Factor Alpha (TNFα) on Endoscopic and Mucosal Healing in Patients Suffering From Active Crohn's Disease.
Brief Title: Mucosal Healing Study in Crohn's Disease (CD)
Acronym: MUSIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C87043; EudraCT Number 2005-003977-25 (Other: EudraCT)
Record Dates: First submitted 2006-02-27; First posted 2006-02-28 (Estimated); Results first posted 2010-01-18 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2011-02

CONDITIONS: Crohn's Disease
Keywords: Certolizumab pegol; Crohn's disease; Mucosal healing
MeSH Terms: conditions — Crohn Disease | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CDP870 400 mg (Experimental): Certolizumab pegol (CDP870) 400 mg
  Interventions: Biological: Certolizumab pegol

INTERVENTIONS:
Biological: Certolizumab pegol — Certolizumab pegol (CDP870) 400 mg administered subcutaneously (sc) at Weeks 0, 2 and 4 (induction doses), then every 4 weeks (Q4W) until Week 52. Investigators can escalate dosage to CDP870 400 mg 2-weekly (Q2W) at any time after Week 10 for lack of response/remission. After Week 52 patients can continue to receive treatment until study drug end, either Q4W or Q2W, according to their administration frequency at Week 52.
  Other Names: Cimzia; CZP; CDP870

SUMMARY:
The aim of the study will be to investigate the effect of certolizumab pegol on the intestinal mucosa in active Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from active Crohn's disease [Crohn's Disease Activity Index(CDAI) ≥ 220 and ≤ 450] and at least 2 segments with endoscopic ulcerative lesions with Baseline Crohn's Disease Endoscopic Index of Severity (CDEIS) ≥ 8
* Patients who need to be treated by anti-tumor necrosis factor (anti-TNF) therapy

Exclusion Criteria:

* Obstructive intestinal strictures, bowel resection, proctocolectomy or total colectomy, current total parenteral nutrition, short bowel syndrome
* History of tuberculosis or positive tests for tuberculosis at screening
* All the concomitant diseases or pathological conditions that could interfere with Crohn's disease assessment or to be harmful for the well being of the patient
* Previous clinical trials and previous biological therapy that could interfere with the results in the present clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2006-02; Primary Completion 2008-01 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (19):
- Belgium (4):
  - Bonheiden
  - Brussels
  - Edegem
  - Leuven
- France (13):
  - Amiens
  - Besançon
  - Chambray-lès-Tours
  - Clichy
  - Grenoble
  - Lille
  - Marseille
  - Nice
  - Paris
  - Reims
  - Rouen
  - Strasbourg
  - Vandœuvre-lès-Nancy
- Germany (2):
  - Berlin
  - Bonn

REFERENCES:
- [Derived] Colombel JF, Sandborn WJ, Allez M, Dupas JL, Dewit O, D'Haens G, Bouhnik Y, Parker G, Pierre-Louis B, Hebuterne X. Association between plasma concentrations of certolizumab pegol and endoscopic outcomes of patients with Crohn's disease. Clin Gastroenterol Hepatol. 2014 Mar;12(3):423-31.e1. doi: 10.1016/j.cgh.2013.10.025. Epub 2013 Nov 1. PMID 24184736
- [Derived] Hebuterne X, Lemann M, Bouhnik Y, Dewit O, Dupas JL, Mross M, D'Haens G, Mitchev K, Ernault E, Vermeire S, Brixi-Benmansour H, Moreels TG, Mary JY, Marteau P, Colombel JF. Endoscopic improvement of mucosal lesions in patients with moderate to severe ileocolonic Crohn's disease following treatment with certolizumab pegol. Gut. 2013 Feb;62(2):201-8. doi: 10.1136/gutjnl-2012-302262. Epub 2012 Apr 23. PMID 22525883
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in sites from Germany, France and Belgium between February 2006 and October 2007. The last patient attended their Week 54 visit in December 2009.
Groups:
- CDP870 400 mg: Certolizumab pegol (CDP870) 400 mg administered at Weeks 0, 2 and 4 (induction doses), then every 4 weeks (Q4W) until Week 52. Investigators can escalate dosage to CDP870 400 mg 2-weekly (Q2W) at any time after Week 10 for lack of response/remission. After Week 52 patients can continue to receive treatment until study drug is approved and available on the market, according to their administration frequency at Week 52 or transition to a standard care regimen or medical need program according to local regulations.
Period: Overall Study
Arm/Group | CDP870 400 mg
Started | 89
Completed | 53
Not Completed | 36
Not completed — Adverse Event | 13
Not completed — Lack of Efficacy | 18
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 3
Not completed — Other: Incompliance | 1

BASELINE CHARACTERISTICS:
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 89
Age, Categorical [Count of Participants; unit: Participants] — Note: The 4 patients in the '<=18 years' category were all 18 years of age at Baseline.
  Participants
    <=18 years | 4
    Between 18 and 65 years | 85
    >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 30.19 (9.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 30
Region of Enrollment [Number; unit: participants]
  France | 68
  Belgium | 16
  Germany | 5

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in CDEIS (Crohn's Disease Endoscopic Index of Severity) Score at Week 10 Using Local Non-blinded Assessments
Description: The CDEIS (Crohn's Disease Endoscopic Index of Severity) score provides a measure of mucosal inflammation. Generally, scores range from 0-30. A higher score indicates more severe mucosal inflammation, thus a negative change from Baseline (i.e., Week 10 score minus Baseline score) indicates improvement.
Time Frame: Baseline, Week 10
Population: Of the 89 patients in the Intent to Treat Population, 78 patients had data at both Baseline and Week 10, and are included in this summary. Change from Baseline has been calculated as the Week 10 score minus the Baseline score, thus a negative Change from Baseline indicates improvement.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 78
score on a scale | -6.47 (5.01) [-7.60 to -5.34]

2. Secondary Outcome: Percentage of Patients Achieving Mucosal Healing at Week 10 Using Local Non-blinded Assessments
Description: Mucosal healing is defined as complete absence of ulceration contribution in the CDEIS (Crohn's Disease Endoscopic Index of Severity) score
Time Frame: Week 10
Population: Of the 89 patients in the Intent to Treat Population, 78 patients had data at Week 10, and are included in this summary. Percentage of patients is calculated by dividing the number of patients who achieved mucosal healing at Week 10 by the total number of patients with data collected, multiplied by 100.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 78
percentage of patients | 5.1 [1.4 to 12.6]

3. Secondary Outcome: Percentage of Patients Achieving Mucosal Healing at Week 10 Using Central Blinded Assessments
Description: as for outcome 2
Time Frame: Week 10
Population: Of the 89 patients in the Intent to Treat Population, 51 patients were in the subpopulation who had a blinded assessment at Week 10 and are included here. Percentage of patients is calculated by dividing the number of patients who achieved mucosal healing at Week 10 by the total number of patients with data collected, multiplied by 100.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 51
percentage of patients | 3.9 [0.5 to 13.5]

4. Secondary Outcome: Percentage of Patients Achieving Mucosal Healing at Week 54 Using Local Non-blinded Assessments
Description: as for outcome 2
Time Frame: Week 54
Population: Of the 89 patients in the Intent to Treat Population, 53 patients had data at Week 54, and are included in this summary. Percentage of patients is calculated by dividing the number of patients who achieved mucosal healing at Week 54 by the total number of patients with data collected, multiplied by 100.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 53
percentage of patients | 13.2 [5.5 to 25.3]

5. Secondary Outcome: Percentage of Patients Achieving Mucosal Healing at Week 54 Using Central Blinded Assessments
Description: as for outcome 2
Time Frame: Week 54
Population: Of the 89 patients in the Intent to Treat Population, 33 patients were in the subpopulation who had a blinded assessment at Week 54 and are included here. Percentage of patients is calculated by dividing the number of patients who achieved mucosal healing at Week 54 by the total number of patients with data collected, multiplied by 100.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 33
percentage of patients | 3.0 [0.1 to 15.8]

6. Secondary Outcome: Percentage of Patients With Endoscopic Response (Crohn's Disease Endoscopic Index of Severity (CDEIS) Decrease From Baseline of More Than 5 Points) at Week 10 Using Local Non-blinded Assessments
Description: The CDEIS (Crohn's Disease Endoscopic Index of Severity) score provides a measure of mucosal inflammation. Generally, scores range from 0-30. A higher score indicates more severe mucosal inflammation.
Time Frame: Baseline, Week 10
Population: Of the 89 patients in the Intent to Treat Population, 78 patients had data at Week 10 and at Baseline, and are included here. Percentage of patients is calculated by dividing the number of patients with a CDEIS decrease of at least 5 points at Week 10 by the number of patients with CDEIS data at both Baseline and Week 10, multiplied by 100.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 78
percentage of patients | 61.5 [49.8 to 72.3]

7. Secondary Outcome: Percentage of Patients With Endoscopic Response (Crohn's Disease Endoscopic Index of Severity (CDEIS) Decrease From Baseline of More Than 5 Points) at Week 10 Using Central Blinded Assessments
Description: as for outcome 6
Time Frame: Baseline, Week 10
Population: Of the 89 patients in the Intent to Treat Population, 44 patients had a blinded assessment at Week 10 and at Baseline, and are included here. Percentage patients is calculated by dividing the number of patients with a CDEIS decrease of at least 5 points at Week 10 by the number of patients with CDEIS data at Baseline and Week 10, multiplied by 100.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 44
percentage of patients | 38.6 [24.4 to 54.5]

8. Secondary Outcome: Percentage of Patients With Endoscopic Response (Crohn's Disease Endoscopic Index of Severity (CDEIS) Decrease From Baseline of More Than 5 Points) at Week 54 Using Local Non-blinded Assessments
Description: as for outcome 6
Time Frame: Baseline, Week 54
Population: Of the 89 patients in the Intent to Treat Population, 53 patients had data at Week 54 and at Baseline, and are included here. Percentage of patients is calculated by dividing the number of patients with a CDEIS decrease of at least 5 points at Week 54 by the number of patients with CDEIS data at both Baseline and Week 54, multiplied by 100.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 53
percentage of patients | 62.3 [47.9 to 75.2]

9. Secondary Outcome: Percentage of Patients With Endoscopic Response (Crohn's Disease Endoscopic Index of Severity (CDEIS) Decrease From Baseline of More Than 5 Points) at Week 54 Using Central Blinded Assessments
Description: as for outcome 6
Time Frame: Baseline, Week 54
Population: Of 89 patients in the Intent to Treat Population 28 had matching nonblinded/blinded assessments and are in the subpopulation with blinded assessment at Week 54 and Baseline. Percentage is calculated by dividing the number patients with CDEIS decrease of at least 5 points at Week 54 by the number with CDEIS at Baseline and Week 54, multiplied by 100
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 28
percentage of patients | 39.3 [21.5 to 59.4]

10. Secondary Outcome: Percentage of Patients With Endoscopic Remission (Crohn's Disease Endoscopic Index of Severity (CDEIS) Score Below 6) at Week 10 Using Local Non-blinded Assessments
Description: as for outcome 6
Time Frame: Week 10
Population: Of the 89 patients in the Intent to Treat Population, 78 patients had data at Week 10, and are included in this summary. Percentage of patients is calculated by dividing the number of patients with a CDEIS score <6 at Week 10 by the total number of patients with CDEIS data at Week 10, multiplied by 100.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 78
percentage of patients | 42.3 [31.2 to 54.0]

11. Primary Outcome: Mean Change From Baseline in CDEIS (Crohn's Disease Endoscopic Index of Severity) Score at Week 10 Using Central Blinded Assessments
Description: as for outcome 1
Time Frame: Baseline, Week 10
Population: Of the 89 patients in the Intent to Treat Population, 44 patients were in the subpopulation with a blinded assessment at Week 10 and Baseline, and are included in this summary. Change from Baseline has been calculated as the Week 10 score minus the Baseline score, thus a negative Change from Baseline indicates improvement.
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 44
Score on a scale | -3.79 [-5.08 to -2.50]

12. Secondary Outcome: Percentage of Patients With Endoscopic Remission (Crohn's Disease Endoscopic Index of Severity (CDEIS) Score Below 6) at Week 10 Using Central Blinded Assessments
Description: as for outcome 6
Time Frame: Week 10
Population: Of the 89 patients in the Intent to Treat Population, 44 patients had a blinded assessment at Week 10 and Baseline, and are included in this summary. Percentage of patients is calculated by dividing the number of patients with a CDEIS score <6 at Week 10 by the total number of patients with CDEIS data at Week 10, multiplied by 100.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 44
percentage of patients | 45.5 [30.4 to 61.2]

13. Secondary Outcome: Percentage of Patients With Endoscopic Remission (Crohn's Disease Endoscopic Index of Severity (CDEIS) Score Below 6) at Week 54 Using Local Non-blinded Assessments
Description: as for outcome 6
Time Frame: Week 54
Population: Of the 89 patients in the Intent to Treat Population, 53 patients had data at Week 54, and are included in this summary. Percentage of patients is calculated by dividing the number of patients with a CDEIS score <6 at Week 54 by the total number of patients with CDEIS data at Week 54, multiplied by 100.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 53
percentage of patients | 28.3 [16.8 to 42.3]

14. Secondary Outcome: Percentage of Patients With Endoscopic Remission (Crohn's Disease Endoscopic Index of Severity (CDEIS) Score Below 6) at Week 54 Using Central Blinded Assessments
Description: as for outcome 6
Time Frame: Week 54
Population: Of 89 patients in the Intent to Treat Population, 28 had matching nonblinded/blinded assessments and were in the subpopulation with a blinded assessment at Week 54 and Baseline. Percentage is calculated by dividing the number of patients with a CDEIS score <6 at Week 54 by the total number of patients with CDEIS data at Week 54, multiplied by 100.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 28
percentage of patients | 32.1 [15.9 to 52.4]

15. Secondary Outcome: Percentage of Patients With Endoscopic Complete Remission (Crohn's Disease Endoscopic Index of Severity (CDEIS) Score Below 3) at Week 10 Using Local Non-blinded Assessments
Description: as for outcome 6
Time Frame: Week 10
Population: Of the 89 patients in the Intent to Treat Population, 78 patients had data at Week 10, and are included in this summary. Percentage of patients is calculated by dividing the number of patients with a CDEIS score <3 at Week 10 by the total number of patients with CDEIS data at Week 10, multiplied by 100.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 78
percentage of patients | 11.5 [5.4 to 20.8]

16. Secondary Outcome: Percentage of Patients With Endoscopic Complete Remission (Crohn's Disease Endoscopic Index of Severity (CDEIS) Score Below 3) at Week 10 Using Central Blinded Assessments
Description: as for outcome 6
Time Frame: Week 10
Population: Of the 89 patients in the Intent to Treat Population, 44 patients had a blinded assessment at Week 10 and Baseline, and are included in this summary. Percentage of patients is calculated by dividing the number of patients with a CDEIS score <3 at Week 10 by the total number of patients with CDEIS data at Week 10, multiplied by 100.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 44
percentage of patients | 20.5 [9.8 to 35.3]

17. Secondary Outcome: Percentage of Patients With Endoscopic Complete Remission (Crohn's Disease Endoscopic Index of Severity (CDEIS) Score Below 3) at Week 54 Using Local Non-blinded Assessments
Description: as for outcome 6
Time Frame: Week 54
Population: Of the 89 patients in the Intent to Treat Population, 53 patients had data at Week 54, and are included in this summary. Percentage of patients is calculated by dividing the number of patients with a CDEIS score <3 at Week 54 by the total number of patients with CDEIS data at Week 54, multiplied by 100.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 53
percentage of patients | 18.9 [9.4 to 32.0]

18. Secondary Outcome: Percentage of Patients With Endoscopic Complete Remission (Crohn's Disease Endoscopic Index of Severity (CDEIS) Score Below 3) at Week 54 Using Central Blinded Assessments
Description: as for outcome 6
Time Frame: Week 54
Population: Of 89 patients in the Intent to Treat Population, 28 had matching nonblinded/blinded assessments and were in the subpopulation with a blinded assessment at Week 54 and Baseline. Percentage is calculated by dividing the number of patients with a CDEIS score <3 at Week 54 by the total number of patients with CDEIS data at Week 54, multiplied by 100.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 28
percentage of patients | 17.9 [6.1 to 36.9]

19. Secondary Outcome: Change From Baseline in Histological Crohn's Disease Score at Week 10 Using Central Blinded Assessment
Description: The histological Crohn's disease score combines active inflammatory changes: infiltration of mononuclear cells, polymorphonuclear cells, presence of erosions and/or ulcers, and chronic architectural changes. Scores range from 0 to 44, with higher scores indicating greater disease.
Time Frame: Baseline, Week 10
Population: Of the 89 patients in the Intent to Treat Population, 75 patients had data at Week 10 and at Baseline for the blinded assessment, and are included in this summary. Change from Baseline has been calculated as the Week 10 score minus the Baseline score, thus a negative change from Baseline indicates improvement.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 75
score on a scale | -1.4 (3.7)

20. Secondary Outcome: Change From Baseline in Histological Crohn's Disease Score at Week 54 Using Central Blinded Assessment
Description: as for outcome 19
Time Frame: Baseline, Week 54
Population: Of the 89 patients in the Intent to Treat Population, 52 patients had data at Week 54 and at Baseline for blinded assessment, and are included in this summary. Change from Baseline has been calculated as the Week 54 score minus the Baseline score, thus a negative Change from Baseline indicates improvement.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 52
score on a scale | -2.5 (4.3)

21. Secondary Outcome: Percentage of Patients Achieving Crohn's Disease Activity Index (CDAI) Response (Defined as a Decrease of at Least 100 Points in CDAI Score From Baseline) at Week 10
Description: Crohn's disease activity index (CDAI) responders are patients achieving clinical response (a reduction in CDAI score of at least 100 points from Baseline). CDAI is used to quantify the symptoms of Crohn's disease. A score of 150 or below indicates remission and a score above 450 indicates extremely severe disease.
Time Frame: Baseline, Week 10
Population: The 89 patients from Intent to Treat Population are included in this summary. In case of missing CDAI score, patients are counted as non-responders. Percentage is calculated by dividing the number of patients with a CDAI decrease of at least 100 points at Week 10 by the total number of patients in the Intent to Treat Population, multiplied by 100.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 89
percentage of patients | 50.6 [39.8 to 61.3]

22. Secondary Outcome: Percentage of Patients Achieving Crohn's Disease Activity Index (CDAI) Response (Defined as a Decrease of at Least 100 Points in CDAI Score From Baseline) at Week 54
Description: as for outcome 21
Time Frame: Baseline, Week 54
Population: The 89 patients from Intent to Treat Population are included in this summary. In case of missing CDAI score, patients are counted as non-responders. Percentage is calculated by dividing the number of patients with a CDAI decrease of at least 100 points at Week 54 by the total number of patients in the Intent to Treat Population, multiplied by 100.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 89
percentage of patients | 32.6 [23.0 to 43.3]

23. Secondary Outcome: Percentage of Patients Achieving Crohn's Disease Activity Index (CDAI) Remission (Defined as a CDAI Score Less Than or Equal to 150) at Week 10
Description: as for outcome 21
Time Frame: Week 10
Population: The 89 patients from Intent to Treat Population are included in this summary. In case of missing CDAI score, patients are counted as remitters. Percentage is calculated by dividing the number of patients with a CDAI less than or equal to 150 points at Week 10 by the total number of patients in the Intent to Treat Population, multiplied by 100.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 89
percentage of patients | 46.1 [35.4 to 57.0]

24. Secondary Outcome: Percentage of Patients Achieving Crohn's Disease Activity Index (CDAI) Remission (Defined as a CDAI Score Less Than or Equal to 150) at Week 54
Description: as for outcome 21
Time Frame: Week 54
Population: The 89 patients from Intent to Treat Population are included in this summary. In case of missing CDAI score, patients are counted as remitters. Percentage is calculated by dividing the number of patients with a CDAI less than or equal to 150 points at Week 54 by the total number of patients in the Intent to Treat Population, multiplied by 100.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 89
percentage of patients | 27.0 [18.1 to 37.4]

25. Secondary Outcome: Geometric Mean C-Reactive Protein (CRP) Level (mg/L) at Week 10
Time Frame: Week 10
Population: Of the 89 patients in the Intent to Treat Population, 76 patients had plasma level data at Week 10 and are included in this summary.
Measure: Geometric Mean (Full Range); unit: mg/L
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 76
mg/L | 6.84 [0.2 to 219.3]

26. Secondary Outcome: Ratio to Baseline of C-Reactive Protein (CRP) Level (mg/L) at Week 10
Description: Ratio is calculated as the Week 10 value divided by the Baseline value for patients with data at both timepoints.
Time Frame: Baseline, Week 10
Population: Of the 89 patients in the Intent to Treat Population, 76 patients had plasma levels taken at Week 10 and Baseline and are included in this summary. Ratio is calculated as the Week 10 value divided by the Baseline value for patients with data at both timepoints.
Measure: Geometric Mean (Full Range); unit: ratio
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 76
ratio | 0.40 [0 to 23.1]

27. Secondary Outcome: Geometric Mean C-Reactive Protein (CRP) Level (mg/L) at Week 52
Time Frame: Week 52
Population: Of the 89 patients in the Intent to Treat Population, 51 patients had plasma level data at Week 54 and are included in this summary.
Measure: Geometric Mean (Full Range); unit: mg/L
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 51
mg/L | 10.24 [0.3 to 99.5]

28. Secondary Outcome: Ratio to Baseline of C-Reactive Protein (CRP) Level (mg/L) at Week 52
Description: The ratio is calculated as the Week 52 value divided by Baseline value for patients with data at both timepoints.
Time Frame: Baseline, Week 52
Population: Of the 89 patients in the Intent to Treat Population, 51 patients had plasma level data at Week 54 and Baseline and are included in this summary. Ratio was calculated by dividing the Week 54 value by the Baseline value for the patients with data at both timepoints.
Measure: Geometric Mean (Full Range); unit: ratio
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 51
ratio | 0.52 [0 to 16.6]

29. Secondary Outcome: Correlation Between Mean C-Reactive Protein (CRP) Plasma Level and Crohn's Disease Activity Index (CDAI) Score at Week 10
Description: as for outcome 21
Time Frame: Week 10
Population: Of the 89 patients in the Intent to Treat Population, 73 patients had plasma level data and a CDAI score at Week 10 and are included in this summary.
Measure: Number (95% Confidence Interval); unit: Pearson Correlation Coefficient
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 73
Pearson Correlation Coefficient | 0.043 [0.000 to 0.270]

30. Secondary Outcome: Correlation Between Mean C-Reactive Protein (CRP) Plasma Level and Crohn's Disease Endoscopic Index of Severity (CDEIS) Score at Week 10 Using Local Non-blinded Assessment
Description: as for outcome 6
Time Frame: Week 10
Population: Of the 89 patients in the Intent to Treat Population, 76 patients had plasma level data and a CDEIS score at Week 10 and are included in this summary.
Measure: Number (95% Confidence Interval); unit: Pearson Correlation Coefficient
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 76
Pearson Correlation Coefficient | 0.131 [0.000 to 0.346]

31. Secondary Outcome: Correlation Between Mean C-Reactive Protein (CRP) Plasma Level and Crohn's Disease Endoscopic Index of Severity (CDEIS) Score at Week 10 Using Central Blinded Assessment
Description: as for outcome 6
Time Frame: Week 10
Population: Of the 89 patients in the Intent to Treat Population, 51 patients were in the subpopulation with a blinded assessment at Week 10. 48 patients had both CDEIS and CRP data at Week 10.
Measure: Number (95% Confidence Interval); unit: Pearson Correlation Coefficient
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 48
Pearson Correlation Coefficient | 0.646 [0.443 to 0.786]

32. Secondary Outcome: Correlation Between Mean C-Reactive Protein (CRP) Plasma Level and Histological Crohn's Disease Score at Week 10 Using Central Blinded Assessment
Description: as for outcome 19
Time Frame: Week 10
Population: Of the 89 patients in the Intent to Treat Population, 72 patients had plasma data and histological Crohn's disease score assessment at Week 10, and are included in this summary.
Measure: Number (95% Confidence Interval); unit: Pearson Correlation Coefficient
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 72
Pearson Correlation Coefficient | 0.086 [0.000 to 0.312]

33. Secondary Outcome: Change From Baseline in Crohn's Disease Endoscopic Index of Severity (CDEIS) Score at Week 54 Using Local Non-blinded Assessment
Description: as for outcome 6
Time Frame: Baseline, Week 54
Population: Of the 89 patients in the Intent to Treat Population, 52 had a CDEIS score at Week 54 and at Baseline and are included here. Change from Baseline has been calculated as the Week 54 score minus the Baseline score, thus a negative Change from Baseline indicates improvement.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 52
score on a scale | -5.49 (7.02)

34. Secondary Outcome: Change From Baseline in Crohn's Disease Endoscopic Index of Severity (CDEIS) Score at Week 54 Using Central Blinded Assessment
Description: as for outcome 6
Time Frame: Baseline, Week 54
Population: Of 89 patients in the Intent to Treat Population, 28 had matching nonblinded/blinded assessments and were in the subpopulation with a blinded assessment at Week 54 and Baseline. Change from Baseline has been calculated as the Week 54 score minus the Baseline score, thus a negative Change from Baseline indicates improvement.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 28
score on a scale | -2.95 (7.13)

35. Secondary Outcome: Change From Baseline in Crohn's Disease Activity Index (CDAI) Score at Week 10
Description: as for outcome 21
Time Frame: Baseline, Week 10
Population: Of the 89 patients in the Intent to Treat Population, 73 patients had data at both Baseline and Week 10, and are included in this summary. Change from Baseline has been calculated as the Week 10 score minus the Baseline score, thus a negative Change from Baseline indicates improvement.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 73
score on a scale | -148.82 (109.61)

36. Secondary Outcome: Change From Baseline in Crohn's Disease Activity Index (CDAI) Score at Week 54
Description: as for outcome 21
Time Frame: Baseline, Week 54
Population: Of the 89 patients in the Intent to Treat Population, 39 had CDAI scores at Week 54 and Baseline and are included in this summary. Change from Baseline has been calculated as the Week 54 score minus the Baseline score, thus a negative Change from Baseline indicates improvement.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CDP870 400 mg
Number analyzed (Participants) | 39
score on a scale | -169.59 (109.98)

ADVERSE EVENTS:
Time Frame: The adverse event summaries are based on data collected during the 54 weeks of the study for all 89 patients.
Arm/Group | CDP870 400 mg
Serious Adverse Events (participants affected / at risk) | 34/89
Other Adverse Events (participants affected / at risk) | 83/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CDP870 400 mg (N=89)
Abdominal abscess (Infections and infestations) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Abdominal wall abscess (Infections and infestations) | 1 (1)
Abdominal wall mass (Gastrointestinal disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Anal abscess (Infections and infestations) | 5 (6)
Anal fistula (Gastrointestinal disorders) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2)
Asthenia (General disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Clostridial infection (Infections and infestations) | 1 (1)
Colitis pseudomembranous (Infections and infestations) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 5 (6)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Enterocutaneous fistula (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Genital abscess (Infections and infestations) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Hyperthermia (General disorders) | 1 (1)
Ileal stenosis (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Keratorhexis (Injury, poisoning and procedural complications) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1)
Localised infection (Infections and infestations) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Perianal abscess (Infections and infestations) | 3 (3)
Perineal abscess (Infections and infestations) | 1 (1)
Perineal fistula (Reproductive system and breast disorders) | 2 (2)
Pregnancy on oral contraceptive (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Serum sickness (Immune system disorders) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CDP870 400 mg (N=89)
Abdominal pain (Gastrointestinal disorders) | 18 (21)
Abdominal pain upper (Gastrointestinal disorders) | 10 (14)
Acne (Skin and subcutaneous tissue disorders) | 9 (9)
Anaemia (Blood and lymphatic system disorders) | 8 (10)
Anal fissure (Gastrointestinal disorders) | 15 (18)
Anal fistula (Gastrointestinal disorders) | 6 (6)
Anxiety (Psychiatric disorders) | 5 (7)
Aphthous stomatitis (Gastrointestinal disorders) | 10 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 27 (43)
Asthenia (General disorders) | 18 (22)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (10)
Bronchitis (Infections and infestations) | 9 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Crohn's disease (Gastrointestinal disorders) | 11 (11)
Diarrhoea (Gastrointestinal disorders) | 13 (20)
Dizziness (Nervous system disorders) | 7 (8)
Dyspepsia (Gastrointestinal disorders) | 6 (7)
Fatigue (General disorders) | 7 (7)
Gastroenteritis (Infections and infestations) | 8 (9)
Haemorrhoids (Gastrointestinal disorders) | 8 (10)
Headache (Nervous system disorders) | 30 (56)
Herpes simplex (Infections and infestations) | 11 (16)
Influenza (Infections and infestations) | 7 (7)
Influenza like illness (General disorders) | 7 (7)
Injection site erythema (General disorders) | 7 (8)
Insomnia (Psychiatric disorders) | 10 (10)
Iron deficiency (Metabolism and nutrition disorders) | 5 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (8)
Nasopharyngitis (Infections and infestations) | 21 (37)
Nausea (Gastrointestinal disorders) | 16 (26)
Night sweats (Skin and subcutaneous tissue disorders) | 5 (5)
Pharyngitis (Infections and infestations) | 11 (12)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 (12)
Proctalgia (Gastrointestinal disorders) | 5 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (7)
Pyrexia (General disorders) | 15 (20)
Rectal haemorrhage (Gastrointestinal disorders) | 5 (5)
Rhinitis (Infections and infestations) | 8 (9)
Sinusitis (Infections and infestations) | 6 (7)
Urinary tract infection (Infections and infestations) | 8 (14)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 6 (6)
Vomiting (Gastrointestinal disorders) | 11 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.